CLINICAL TRIAL: NCT03360526
Title: What is the Best Sperm Source and Way of Sperm Selection in Cases With Abnormal Static Oxidation Reduction Potential (sORP) Levels on the Day of ICSI?
Brief Title: What is the Best Sperm Source and Way of Sperm Selection in Cases With Abnormal sORP Levels on the Day of ICSI?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ganin Fertility Center (Other)
Collaborators: The Cleveland Clinic (Other); University of the Western Cape (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMSH25390
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Oxidative Stress
Keywords: PICSI; ORP; TESA; seminal oxidation reduction potential

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICSI (Active Comparator): Physiological ICSI
  Interventions: Device: PICSI
- TESA (Experimental): Testicular sperm aspiration
  Interventions: Procedure: TESA

INTERVENTIONS:
Device: PICSI — Semen processing is done by double layer density gradient method followed by adding Sperm to the dot of hyaluronan on the PICSI dish, within minutes the bound sperm are attached by their acrosome to the surface of the dot. (Selecting an individual bound sperm with enhanced genetic and developmental integrity ensures that the sperm selected is the optimal sperm from the sample for oocyte injection.
  Arms: PICSI
Procedure: TESA — Patients will undergo TESA which is performed by sticking a needle in the testis and aspirating fluid and tissue with negative pressure then examine the sample for presence of motile
  sperms followed by sample processing and oocyte injection.
  Arms: TESA

SUMMARY:
Does the level of statistic oxidation reduction potential (sORP) affects the choice of sperm source or sperm selection method used during ICSI.

DETAILED DESCRIPTION:
Reactive oxygen species (ROS) are an integral component of sperm developmental physiology, capacitation, and function. Elevated ROS levels, from processes such as infection or inflammation, can be associated with male infertility and also decreases the overall ICSI success rates[1][2]

Several techniques are available for measuring ROS, but only Mioxsys can measure the imbalance between production of reactive oxygen species (ROS) and activity of the antioxidant defense system in semen in terms of sORP. Mioxsys is a robust test that gives the result in a very short time, so it became applicable to test sORP on day of ICSI [2]

Injection with sperm selected by PICSI dishes or testicular sperm aspiration (TESA) is thought to decrease or eliminate the unwanted ROS but none of them was reported to be more efficient than the other with regards to the clinical outcomes.

A sperm selection technique based on sperm membrane binding to hyaluronic acid (PICSI Dish), the main substrate of the oocyte zona pellucida, could improve the likelihood of obtaining better sperm for ICSI. It is thought that excessive ROS damages sperm membranes, reduces sperm motility, and induces sperm DNA damage [3]

The topographic assessment of sperm chromatin integrity throughout the male genital tract suggested that there is a disruption in DNA packing during spermiogenesis that does not allow sperm chromatin to withstand oxidative stressors, possibly compounded by a compromised total antioxidant capacity in the seminal fluid [4]. The utilization of testicular spermatozoa may represent a viable option for men with high ROS level in their ejaculates.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of abnormal male semen parameters such as abnormal sperm parameters according to WHO 2010 or high DNA fragmentation using TUNEL as a cause of couple infertility.
* Abnormal sORP level on the day of ICSI.
* Males with mild OTA (oligoteratoasthenozoospermia).
* Female aged 18-35 years.
* Normo responder ( > 8 mature oocytes)
* Male will have to refrain from ejaculation no less than 1 day but no greater than 3 days prior semen specimen production on day of oocyte retrieval

Exclusion Criteria:

* Normal Semen fluid analysis ( WHO 2010) during the initial assessment of the male
* Normal sORP levelat the day of ICSI
* Leukocytospermia
* Presence of varicocele.
* Known genetic abnormality
* Use of sperm donation or cryopreserved sperm
* Use of Oocyte donation
* Use of gestational carrier
* Presence of any of the endometrial factors that affect embryo implantation such as hydrosalpings, adenomyosis or previously known uterine infection
* Any contradictions to undergoing in vitro fertilization or gonadotropin stimulation

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male Since Born
Enrollment: 820 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 20 weeks of gestation
  Defined as the proportion of pregnancies that had completed ≥20 weeks of gestation.

SECONDARY OUTCOMES:
Fertilization rate | 16-18 hours
  Defined as the proportion of 2PNs formed over the injected oocytes
Cleavage rate | 3 days
  Defined as the proportion of cleaved embryos on day 3 over the injected oocytes
Blastulation rate | 5-6 days
  Defined as the proportion of blastocysts formed on day 5 or 6 over the cleaved embryos on day 3
Blastocyst quality rate | 5-6 days
  Defined as the assessment of blastocyst quality according to Gardner's criteria into: good, fair or bad in terms of percentage of the total formed blastocysts
Pregnancy rate | 14 days following embryo transfer
  Defined as clinical pregnancy per embryo(s) transfer
Implantation rate | 6- 8 weeks following embryo transfer]
  Defined as number of gestational sacs with fetal heart beat, shown by ultrasound in gestational week 6 over number of embryo(s) transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Hasanen, BSc, Principal Investigator — Ganin Fertility Center, Cairo, Egypt; Hosam Zaki, MSc, FRCOG, Study Chair — Ganin Fertility Center, Cairo, Egypt; Khaled Elqusi, BSc, Principal Investigator — Ganin Fertility Center, Cairo, Egypt; Ashok Agarwal, Ph.D, Study Director — American Center of reproductive medicine, Cleveland Clinic, Ohio, USA; Ralph Henkel, PhD, Principal Investigator — University of the Western Cape; Hanaa Elkhedr, ABB( ELD), Principal Investigator — Ganin Fertility Center, Cairo, Egypt
Locations (1):
- Ganin Fertility center, Maadi, Cairo Governorate, Egypt

REFERENCES:
- [Background] Agarwal A, Sharma R, Roychoudhury S, Du Plessis S, Sabanegh E. MiOXSYS: a novel method of measuring oxidation reduction potential in semen and seminal plasma. Fertil Steril. 2016 Sep 1;106(3):566-573.e10. doi: 10.1016/j.fertnstert.2016.05.013. Epub 2016 May 31. PMID 27260688
- [Background] Agarwal A, Roychoudhury S, Sharma R, Gupta S, Majzoub A, Sabanegh E. Diagnostic application of oxidation-reduction potential assay for measurement of oxidative stress: clinical utility in male factor infertility. Reprod Biomed Online. 2017 Jan;34(1):48-57. doi: 10.1016/j.rbmo.2016.10.008. Epub 2016 Oct 20. PMID 27839743
- [Background] Natali A, Turek PJ. An assessment of new sperm tests for male infertility. Urology. 2011 May;77(5):1027-34. doi: 10.1016/j.urology.2010.10.005. Epub 2011 Jan 22. PMID 21256575
- [Background] T. Cozzubbo, Q.V. Neri, M. Goldstein, Z. Rosenwaks, G.D. Palermo. Topographic mapping of sperm DNA fragmentation within the male genital tract.